CLINICAL TRIAL: NCT06729619
Title: Concentration Monitoring of Anti-infective Drugs in Human Cerebrospinal Fluid and Its Clinical Application
Status: Active, not recruiting | Type: Observational
Sponsor: Xueyan Cui (Other)
Responsible Party: Sponsor-Investigator, Xueyan Cui, associate professor of pharmacy, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: QFS-CXY-2023-ZSGR-001
Record Dates: First submitted 2024-12-04; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Intracranial Infection; Central Infection
Keywords: Intracranial infection; Cerebrospinal fluid concentration; Anti-infective drugs
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with central infection
  Interventions: Drug: The concentration of anti-infective drugs in blood and cerebrospinal fluid will be determined.

INTERVENTIONS:
Drug: The concentration of anti-infective drugs in blood and cerebrospinal fluid will be determined. — Blood and cerebrospinal fluid concentrations of anti-infective drugs such as vancomycin, meropenem, linezolid, cefoperazone sulbactam and ceftazidime ababactam will be monitored after the drug reaches a steady state.

SUMMARY:
At least 50 patients with intracranial infection receiving anti-infective drugs such as vancomycin, meropenem, linezolid, cefoperazone sulbactam, ceftazidime and avibactam were included in each group for pharmacokinetic study, and the outcomes and adverse events of intracranial infection treatment were observed.

DETAILED DESCRIPTION:
This study intends to establish a high performance liquid phase method to determine the concentration of anti-infective drugs such as vancomycin, meropenem, linezolid, cefoperazone sulbactam, ceftazidime abvibactam and other anti-infective drugs in cerebrospinal fluid, determine the concentration of cerebrospinal fluid in patients with central infection, and simultaneously determine the concentration of blood drugs at the same time point, optimize the clinical treatment plan by combining the concentration of cerebrospinal fluid and blood drugs, and explore the optimal concentration range of cerebrospinal fluid. At the same time, it can improve the cure rate of central infection, shorten the course of treatment and reduce the occurrence of adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. clinically diagnosed as central infection (cerebrospinal fluid culture is positive with clinical infection symptoms) or suspected as central infection (abnormal cerebrospinal fluid examination, such as hypoglycemia, < 50%; High protein, > 50 mg/dl; The number of cells increased with clinical infection symptoms, but no cerebrospinal fluid culture was positive)
3. receiving anti-infection treatment such as vancomycin or meropenem or linezolid or cefoperazone sulbactam;
4. Sign the informed consent form.

Exclusion Criteria:

1. There is no cerebrospinal fluid to determine the concentration;
2. allergic to drugs;
3. Other factors that researchers think are not suitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample size of patients with central infection was collected from November 2023 to the completion.
  Recruitment location: First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital, Shandong Province).
  Research time: 2023-2026.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cerebrospinal fluid concentration of anti-infective drugs | 2023-2026
  We will establish a methodology for determining the concentrations of anti-infective drugs such as vancomycin, meropenem, linezolid, cefoperazone sulbactam and ceftazidime ababactam in cerebrospinal fluid by high performance liquid chromatography, and determine the drug concentrations in cerebrospinal fluid of patients with central infection, and simultaneously determine the blood drug concentrations at the same time point.

SECONDARY OUTCOMES:
The incidence of adverse events caused by treatment | 2023-2026
  In a clinical trial, the probability of an unexpected and adverse medical event that occurs after a patient or clinical subject receives a trial drug, but it does not necessarily have a causal relationship with the treatment.
Treatment outcome of central infection | 2023-2026
  If there are blood routine tests, cerebrospinal fluid tests and procalcitonin tests before and after drug treatment, relevant information, combined drugs and adverse events will be collected to evaluate the effectiveness and safety of drug treatment for central infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Provincial Qianfoshan Hospital, Jinan, Shandong Provincial, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF